CLINICAL TRIAL: NCT06556212
Title: Real-time Feedback in Swimming: Workout Compliance and Swimming Performance Outcomes Using Smart Swim Goggles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Simon Fraser University (Other)
Collaborators: Form Athletica Inc. (Unknown)
Responsible Party: Principal Investigator, David Clarke, Associate Professor, Simon Fraser University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 30001408
Record Dates: First submitted 2024-08-10; First posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Effect of Real-time Visual Feedback on Participant Compliance, Motivation, and Performance in Swimming
Keywords: feedback, sensory; feedback, physiological; swimming; physical fitness

STUDY DESIGN:
Intervention Model Description: The intervention group ("feedback") will differ from the control group ("non-feedback") in that they will have the FORM goggles display on and receive real-time metrics and guided workouts throughout the remainder of the study. "Non-feedback" will have the display turned on but will only have the workout timer visible during rest. Each group will be provided with the same twelve-week training program that differs only in the prescribed pace for each workout.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Feedback (Experimental): This arm will have the smart swim goggles display on and receive real-time metrics and guided workouts via the goggles throughout the study training period.
  Interventions: Other: Real-time feedback using smart swim goggles
- Non-feedback (No Intervention): This arm will have the smart swim goggles display turned on but will only have the workout timer visible during rest. They will not receive real-time metrics or guided workouts via the goggles.

INTERVENTIONS:
Other: Real-time feedback using smart swim goggles — Smart swim goggles (Form Athletica Inc.) with activity metrics (such as heart rate, swimming pace, and workout instructions) displayed in real-time during a swimming activity.
  Arms: Feedback

SUMMARY:
In August of 2019 a Canadian company, Form Athletica Inc. (FORM), introduced a pair of Smart swimming goggles (FORM goggles) with a built-in see-through display. The FORM Smart Swim Goggles both track and display the following performance metrics in real time: lap time splits, distance, stroke rate, stroke count, distance per stroke, pace, auto-rest, and heart rate. The goggles are also capable of showing structured workouts from inside the goggles. To assess the FORM goggles heart rate monitor, swimmer workout compliance, and swimmer performance adaptations, a group of recreational swimmers will complete familiarization sessions using the FORM goggles, perform a baseline performance test, follow a 12-week training program, and complete a final performance test.

DETAILED DESCRIPTION:
The following research questions guide the study design:

1. Do recreational swimmers exhibit greater workout adherence when utilizing FORM goggles for real-time visual feedback in comparison to recreational swimmers who do not utilize such feedback?
2. Will the utilization of real-time visual feedback lead to higher motivation levels for recreational swimmers in comparison to recreational swimmers who do not utilize such real-time feedback?
3. Will there be a more pronounced performance enhancement among recreational swimmers who employ real-time visual feedback during a 12-week training period, as opposed to recreational swimmers who do not utilize such feedback?

The experiment will be conducted over 13 weeks. Week 1 and the final day of week 13 will be in-person. The remaining weeks/days will be completed by the participants on their own. The in-person days will be carried out in a designated 25-meter indoor swimming pool using 6 lanes with a total of 12 swimmers per session. Video footage will be captured on all in-person days as a reference for any discrepancies in the FORM goggles output, and as a more precise method of measuring the performance test. FORM goggles will be used by all participants.

Prior to Week 1, educational material and the Get Active Questionnaire will be provided to participants. The educational material will include information on standard swimming workout language, session rating of perceived exertion (sRPE), using the FORM goggles, and using the FORM Swim application on a cellular phone. The Get Active Questionnaire will need to be completed prior to commencing testing.

Week 1 sessions will be utilized for familiarization/testing purposes and for recording data for the heart rate validation component of the study. Within each session, all participants will be equipped with an external heart rate monitor (Polar Verity) and 4 will be equipped with an additional heart rate monitor (Garmin HRM-Swim). Two sessions will be designated for the participants to get accustomed to the FORM goggles (face fit, field of view, and user interface). These sessions will consist of standardized workouts between 1000m and 2000m. The remaining session will be used to complete a performance test as described in the paragraph below. Before the data collection commences the following will occur:

* Establishing the participants' understanding of the educational material distributed prior to week 1
* Retrieval of completed Get Active Questionnaires
* Briefing the participants on using the FORM goggles and FORM app by the research personnel

Week 1 will contain a baseline performance test. This performance test will determine the participants' critical swim speed (CSS) through two maximal efforts (400 m front crawl, followed by 50 m front crawl) with adequate rest between to produce "best-effort" swims. At the end of week 1, participants will be stratified and randomized into an intervention group ("feedback") and control group ("non-feedback") and reported using the CONSORT guidelines. "Feedback" will differ from "non-feedback" in that they will have the FORM goggles display on and receive real-time metrics and guided workouts throughout the remainder of the study. "non-feedback" will have the display turned on but will only have the workout timer visible during rest. Each group will be provided with the same twelve-week training program. Within each group there will be three training plan volumes (High, Medium, Low) that participants will be assigned to, ensuring appropriate training load prescription per participant. A swim coach will make the assignments using information from the participants' previous swimming experience, and the participants' baseline CSS. "Feedback" will have the convenience of guided workouts in the FORM goggles, while "non-feedback" will be required to use other methods of remembering their workouts (i.e., paper, standard training application, etc.).

Weeks 2-13 will consist of unsupervised sessions to assess the impact of motivation, compliance and workout adherence on CSS performance. The participants will complete three workouts per week on their own time at their local indoor pool.

Week 13 will conclude with a final CSS performance test on the final workout day.

Workout instructions will be provided via email and in-app to all participants at the beginning of each training week. A questionnaire will be delivered to each participant after each training session to record data such as their perceived effort of the training session, exercise motivation, and exercise enjoyment. An additional questionnaire will be provided every 4 weeks to assess participants' experience with the usability and legibility of the FORM goggles or other utilized workout instruction/performance feedback device.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Can swim 400m front crawl (FR) continuously at a maximum effort
* Can swim a minimum of 3 times a week
* Can swim a minimum of 2000m in a session
* Are not currently injured and have had a minimum of 6 weeks recovery from a previous injury
* Are proficient in FR, backstroke (BK), breaststroke (BR)
* Prepared to dedicate 1-1.5 hours a session for 4 in-person sessions
* Are able to complete 3 workouts a week for 12 weeks on their own on separate days with at least one day in between workouts
* Live in British Columbia, Canada and live max 15km from nearest public pool
* Must be willing to minimize all other forms of physical training during the study period

Exclusion Criteria:

* Current competitive swimmer
* Currently training on a swim team or in a swim club

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2023-03-27 (Actual); Primary Completion 2023-12-09 (Actual); Study Completion 2023-12-09 (Actual)

PRIMARY OUTCOMES:
Compliance: Workout pool length count difference | From Week 2 of the study to the end of Week 13 (Weeks 1 to 12 of the training program).
  Measured as the difference (count) between prescribed pool lengths and completed pool lengths per workout.
Compliance: Interval rest time difference | From Week 2 of the study to the end of Week 13 (Weeks 1 to 12 of the training program).
  Measured as the difference (seconds) between prescribed rest time and actual rest time per rest interval.
Compliance: Interval stroke type difference | From Week 2 of the study to the end of Week 13 (Weeks 1 to 12 of the training program).
  Measured as a "success" (1) or "failure" (0) to complete the prescribed stroke type per swim interval.
Compliance: Interval effort difference | From Week 2 of the study to the end of Week 13 (Weeks 1 to 12 of the training program).
  Measured as a "success" (1) or "failure" (0) to meet the prescribed effort (based on a participant-specific percentage of critical swim speed) per freestyle swim interval.
Compliance: Workout effort difference | From Week 2 of the study to the end of Week 13 (Weeks 1 to 12 of the training program).
  Measured as the difference (count) between prescribed workout effort and participant provided workout effort. Workout effort is quantified using session rating of perceived exertion (sRPE) which is evaluated using the Borg Category-Ratio 10 scale. The minimum value is 0 (indicating no exertion at all) and the maximum value is 10 (indicating maximal exertion).
Motivation: Completed workout difference | From Week 2 of the study to the end of Week 13 (Weeks 1 to 12 of the training program).
  Measured as the difference (count) between prescribed workouts and completed workouts.
Motivation: Questionnaire | From Week 2 of the study to the end of Week 13 (Weeks 1 to 12 of the training program).
  Evaluated after every workout (via an online questionnaire) on a 5-point Likert scale (1 = Strongly Disagree, 5 = Strongly Agree) for the following questions:
  * Accomplishment - "I feel a sense of accomplishment after completing my swim workout"
  * Enjoyment - "I enjoyed my swim workout today"
  * Motivation - "I am motivated to complete my next swim workout"
  Higher scores indicate higher motivation levels.
Performance: Adaptation (Critical swim speed) | From the start of Week 1 of the training program to the end of week 12 of the training program.
  Performance is measured as the difference (metres/second) between the baseline critical swim speed, measured at the end of Week 1 of the study, and the post-training critical swim speed, measured at the end of Week 13 of the study (end of Week 12 of the training program).

SECONDARY OUTCOMES:
Validity: Heart rate sensor | Week 1 of the study
  Is the smart swim goggles integrated photoplethysmography heart rate sensor valid and reliable when compared to an electrocardiogram sensor (Garmin HRM-Swim)?
  Validity will be measured as the difference (beats per minute) between heart rate values from the Garmin HRM-Swim monitor and heart rate values from the smart swim goggles from two separate workouts in Week 1 of the study.

CONTACTS AND LOCATIONS:
Overall Officials: David C Clarke, PhD, Principal Investigator — Simon Fraser University
Locations (1):
- St. George's Senior School, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No